CLINICAL TRIAL: NCT02946476
Title: Prevalence and Prognostic Impact of Noncardiac Comorbidities in Heart Failure Outpatients With Preserved and Reduced Ejection Fraction: A Community-Based Study
Brief Title: Prognostic Impact of Noncardiac Comorbidities in Heart Failure Patients
Acronym: NCC-HF
Status: Completed | Type: Observational
Sponsor: Ospedale Maggiore Di Trieste (Other)
Responsible Party: Principal Investigator, Annamaria Iorio, Principal Investigator, Ospedale Maggiore Di Trieste
Other Study IDs: OMTrieste
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure, Diastolic; Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HFrEF: patients with heart failure and reduced ejection fraction
  Interventions: Other: prognostic impact of non cardiac comorbidities
- HFpEF: patients with heart failure and preserved ejection fraction
  Interventions: Other: prognostic impact of non cardiac comorbidities

INTERVENTIONS:
Other: prognostic impact of non cardiac comorbidities

SUMMARY:
To better understand the public health prognostic impact of noncardiac chronic illnesses, we explored the attributable risk of noncardiac comorbidities on outcomes between heart failure patients with reduced ejection fraction (HFREF) and heart failure patients with preserved ejection fraction (HFpEF) in a large contemporary heart failure (HF) population The adjusted hazard ratio (HR) and the population attributable risk were used to compare the contributions of 15 noncardiac comorbidities to adverse outcome. The comorbidities that contributed to high attributable risk were: anemia, chronic kidney disease, chronic obstructive pulmonary disease, diabetes mellitus, and peripheral artery disease. These findings were similar for HFrEF and HFpEF groups. Interaction analysis confirmed similar results.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive heart failure patients with left ventricular ejction fraction available before or within 3 months from the index visit

Exclusion Criteria:

* We excluded all patients who had severe primary left-sided valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We studied all consecutive heart failure patients with diagnostic codes presenting clinical findings compatible with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 2314 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
overall mortality | 2 years

SECONDARY OUTCOMES:
First all-cause hospitalization | 2 years
Heart Failure hospitalization | 2 years
noncardiovascular hospitalization | 2 years